CLINICAL TRIAL: NCT06308536
Title: Study on the Effect of Concentrated Growth Factor in Promoting the Regeneration and Preservation of Soft and Hard Tissues
Brief Title: Application of Concentrated Growth Factors in Alveolar Ridge Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2023-045
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alveolar Ridge Preservation; Concentrated Growth Factor
Keywords: extraction site preservation; concentrated growth factor; CGF; soft and hard tissue regeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- bone powder + collagen membrane (Active Comparator): Fill the extraction socket with bone powder, and cover the extraction wound with collagen membrane.
  Interventions: Procedure: bone powder + collagen membrane
- bone powder + collagen membrane + CGF membrane (Experimental): Fill the extraction socket with bone powder, and cover the extraction wound with collagen membrane and CGF membrane.
  Interventions: Procedure: bone powder + collagen membrane + CGF membrane
- bone powder mixed wih CGF gel + collagen membrane + CGF membrane (Experimental): Fill the extraction socket with bone powder mixed with CGF gel, and cover the extraction wound with collagen membrane and CGF membrane.
  Interventions: Procedure: bone powder mixed wih CGF gel + collagen membrane + CGF membrane
- bone powder + CGF membrane (Experimental): Fill the extraction socket with bone powder, and cover the extraction wound with CGF membrane.
  Interventions: Procedure: bone powder + CGF membrane

INTERVENTIONS:
Procedure: bone powder + collagen membrane — Fill the extraction socket with Bio-Oss® bone powder, and cover the extraction wound with Bio-Gide® collagen membrane.
  Arms: bone powder + collagen membrane
Procedure: bone powder + collagen membrane + CGF membrane — Fill the extraction socket with Bio-Oss® bone powder, and cover the extraction wound with Bio-Gide® collagen membrane plus CGF membrane(CGF gel is pressed into a film)
  Arms: bone powder + collagen membrane + CGF membrane
Procedure: bone powder mixed wih CGF gel + collagen membrane + CGF membrane — Fill the extraction socket with Bio-Oss® bone powder mixed with CGF gel (CGF gel is cutted into granules ), and cover the extraction wound with Bio-Gide® collagen membrane plus CGF membrane(CGF gel is pressed into a film)
  Arms: bone powder mixed wih CGF gel + collagen membrane + CGF membrane
Procedure: bone powder + CGF membrane — Fill the extraction socket with Bio-Oss® bone powder and cover the extraction wound with CGF membrane(CGF gel is pressed into a film)
  Arms: bone powder + CGF membrane

SUMMARY:
To explore the role of CGF in the regeneration or preservation of soft and hard tissues during tooth extraction site preservation surgery.

DETAILED DESCRIPTION:
A prospective, randomized controlled trial is designed to explore the role of CGF in the regeneration or preservation of soft and hard tissues in extraction site preservation. Using random number table, 20 patients were randomly divided into 4 groups using different filling materials in the extraction socket and materials for the wound sealing. Group A (5cases): bone powder + collagen membrane; Group B (5 cases): bone powder + collagen membrane + CGF membrane; Group C (5 cases): bone powder mixed CGF gel + collagen membrane + CGF membrane; Group D (5 cases): bone powder + CGF membrane.

Extraction and site preservation surgery were performed by the same physician and clinical follow-up was more than 6 months after surgery. The four groups will be compared on several variables, including the changes in pain score, Landry wound healing index, membrane exposure area, keratinized gingival width, buccolingual gingival width, alveolar crest width and height.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily participate in this trial and sign a written informed consent; Patients aged 25 ≤ age ≤ 45 years; The combination of intraoral and imaging examinations confirms that the affected tooth has no preservation value, requires tooth extraction, and the patient is willing to use site preservation; No progressive periodontal disease or acute apical periodontitis in the affected teeth; No long-term history of oral bisphosphonates; Non smoking patients； No systemic diseases such as diabetes and hypertension.

Exclusion Criteria:

Patients who have difficulty tolerating surgery; Patients under 25 years old or above 45 years old; The whole body is accompanied by hypertension, diabetes and other serious systemic diseases, which need to be controlled by drugs; Patients who take oral medication that affects bone metabolism for at least one month due to the need for disease treatment; Patients who take medication that may affect platelet function was used within 3 months due to the need for disease treatment; Patients unable to undergo X-ray imaging examination due to pregnancy or preparation after site preservation surgery; Patients who Smoke; The apical and periodontal inflammation is in the acute phase (purulent phase) Regular follow-up or follow-up for more than 6 months is not allowed

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
the width of keratinized gingiva | preoperative, 3 months and 6 months after surgery
  the width of keratinized gingiva measured by periodontal probe
the horizontal width (from buccal to lingual at the alveolar top ) of gingiva | immediate , 3 months and 6 months postoperative
  the horizontal width of gingiva measured by periodontal probe
the horizontal bone resorption of alveolar crest | immediate , 3 months and 6 months postoperative
  Compared with immediate postoperative, the horizontal width of alveolar crest decreased at 3months and 6 months, postoperative alveolar bone resorption progressed with time
the vertical bone resorption of alveolar crest | immediate , 3 months and 6 months postoperative
  the vertical width of alveolar crest decreased at 3months and 6 months postoperative compared with the immediate postoperative
the average gray value of alveolar bone | immediate , 3 months and 6 months postoperative
  the average gray value of alveolar bone

SECONDARY OUTCOMES:
Landry wound healing index | 7 days and 12 days after surgery
  scores:1,2,3,4,5 according to the gingival healing status
reduction in membrane exposure area | 7 days,12 days and one month after surgery
  membrane exposure area reduce different in four groups
pain score | 1day, 3days after surgerys
  scores: 2,4,6,8,10 using the Wong-Baker facial pain scale revision (FPS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Genying Zhuang, Master, Study Director — The Fourth Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang Procince, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li S, Yang H, Duan Q, Bao H, Li A, Li W, Chen J, He Y. A comparative study of the effects of platelet-rich fibrin, concentrated growth factor and platelet-poor plasma on the healing of tooth extraction sockets in rabbits. BMC Oral Health. 2022 Mar 23;22(1):87. doi: 10.1186/s12903-022-02126-0. PMID 35321697
- [Result] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303